CLINICAL TRIAL: NCT00965653
Title: Open-label, Multicenter, Randomized, Parallel Study to Investigate pk, pd, Efficacy and Safety of Tocilizumab (TCZ, RO4877533) Following Subcutaneous Administration of TCZ 162 mg Weekly or Every Other Week in Combination With Methotrexate in Patients With Rheumatoid Arthritis
Brief Title: A Study of Subcutaneously Administered Tocilizumab in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP22623; 2009-011349-18
Record Dates: First submitted 2009-08-18; First posted 2009-08-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Folic Acid; Methotrexate; tocilizumab

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: folic acid; Drug: methotrexate; Drug: tocilizumab [RoActemra/Actemra]
- 2 (Active Comparator)
  Interventions: Drug: folic acid; Drug: methotrexate; Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: folic acid — >/= 5 mg po weekly
Drug: methotrexate — 7.5 - 25 mg weekly (oral or parenteral)
Drug: tocilizumab [RoActemra/Actemra] — 162 mg sc weekly (QW)for 12 weeks
  Arms: 1
Drug: tocilizumab [RoActemra/Actemra] — 162 mg sc every other week (Q2W) for 12 weeks
  Arms: 2

SUMMARY:
This open-label randomized 2arm study will investigate the pharmacokinetics, pharmacodynamics, efficacy and safety of subcutaneously administered tocilizumab in patients with rheumatoid arthritis who have shown an inadequate response to methotrexate. Patients will be randomized to receive tocilizumab 162 mg sc either weekly or every other week, in combination with methotrexate, for 12 weeks. Assessments will be made at regular intervals during treatment and on the 3 weeks of follow-up.Target sample size is < 50 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 - 75 years of age
* active rheumatoid arthritis of >/= 6 months duration
* inadequate response to at least 12 weeks of methotrexate, the last 8 prior to baseline on stable dose
* swollen joint count (SJC)>/=4, tender joint count (TJC)>/=6 at screening and baseline
* DMARDs and anti-TNFs, other than methotrexate, withdrawn prior to baseline
* oral corticosteroids (</= 10mg/day prednisone or equivalent) and NSAIDS on stable dose </= 4 weeks prior to baseline

Exclusion Criteria:

* rheumatic autoimmune disease other than rheumatoid arthritis
* prior history or current inflammatory joint disease other than rheumatoid arthritis
* major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following enrollment
* functional class IV by ACR classification

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-08; Study Completion 2011-07

PRIMARY OUTCOMES:
Pharmacokinetics of TCZ after QW or Q2W sc administration | multiple sampling after 1st and last dose, weeks 1 and 12, at bi-weekly intervals during treatment and twice on follow-up
Pharmacodynamic responses of CRP | sampling in weeks 1 and 2 and at weekly or bi-weekly intervals throughout treatment
Safety and tolerability, including injection site reaction | laboratory assessments every 2nd week on treatment and after 3 weeks follow-up, injection site evaluation after 1st, 2nd and last injection.

SECONDARY OUTCOMES:
Efficacy according to ACR and DAS-EULAR parameters | assessments on day 1 of weeks 1, 4, 8 and 12
PD responses of IL-6, sIL-6R and anti TCZ antibody | multiple sampling after 1st and last dose, weeks 1 and 12, at bi-weekly intervals during treatment and twice on follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- Canada (3):
  - St. John's, Newfoundland and Labrador
  - Kitchener, Ontario
  - Trois-Rivières, Quebec
- Christchurch, New Zealand
- Spain (3):
  - A Coruña, La Coruña
  - Santiago de Compostela, La Coruña
  - Seville, Sevilla